CLINICAL TRIAL: NCT00931229
Title: Incidence of Hepatitis B Reactivation in Non-Hodgkin's Lymphoma Patients Who Receive Rituximab-containing Chemotherapy and Are Previously Infected With Hepatitis B Virus
Brief Title: Incidence of Hepatitis B Reactivation in Non-Hodgkin's Lymphoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); China Medical University Hospital (Other); Chi Mei Medical Hospital (Other); Taichung Veterans General Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: T1408
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2011-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: hepatitis B reactivation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- entecavir (Experimental): All eligible patients will receive rituximab-CHOP (cyclophosphamide, doxorubicin, vincristine, prednisolone) chemotherapy according to current treatment guidelines.
  Interventions: Drug: entecavir

INTERVENTIONS:
Drug: entecavir — All eligible patients will receive rituximab-CHOP (cyclophosphamide, doxorubicin, vincristine, prednisolone) chemotherapy according to current treatment guidelines. The primary endpoint of this study is the incidence of HBV reactivation, defined by a greater than 10-fold increase, compared with previous nadir levels, of HBV DNA during rituximab-CHOP chemotherapy and within 1 year after completion of the last course of rituximab-CHOP chemotherapy. Patients who have HBV reactivation during the study period will receive free entecavir treatment, one of the standard treatment for chronic hepatitis B, for 48 weeks.

SUMMARY:
This is a single-arm study. Key eligibility criteria include (1) newly diagnosed, diffuse large B-cell or follicular cell non-Hodgkin's lymphoma; (2) negative test for hepatitis B surface antigen (HBsAg) and positive for antibody to hepatitis B core antigen (anti-HBc); (3) adequate bone marrow, liver, and kidney function. All eligible patients will receive rituximab-CHOP (cyclophosphamide, doxorubicin, vincristine, prednisolone) chemotherapy according to current treatment guidelines. The primary endpoint of this study is the incidence of hepatitis B virus (HBV) reactivation, defined by a greater than 10-fold increase, compared with previous nadir levels, of HBV DNA during rituximab-CHOP chemotherapy and within 1 year after completion of the last course of rituximab-CHOP chemotherapy. Patients who have HBV reactivation during the study period will receive free entecavir treatment, one of the standard treatment for chronic hepatitis B, for 48 weeks. The secondary endpoints include the incidence of hepatitis flare, defined as a greater than 3 fold increase of serum alanine aminotransferase (ALT) level that exceeded 100 IU/L, and the efficacy and safety of rituximab-CHOP chemotherapy.

In the T1408 study we enrolled patients with newly diagnosed lymphoma who were HBsAg (-) and anti-HBc (+) and were to receive rituximab-CHOP (cyclophosphamide, doxorubicin, vincristine, prednisolone)-based chemotherapy. Key findings of this study included (1) HBV reactivation, defined as a greater than 10-fold increase in HBV DNA compared with previous nadir levels, occurred to 10-20% of patients, depending on the sensitivity of the HBV DNA tests; (2) no HBV-related death with the prompt anti-viral therapy upon HBV reactivation; (3) patients with HBV reactivation were associated with poorer progression-free survival and overall survival; (4) serological breakthrough (i.e., re-appearance of HBsAg) is an important predictor of HBV-related hepatitis flare.

In this amendment we will enroll more patients to clarify the above findings: (1) the association between HBV reactivation and survival; (2) diagnostic value of quantitative HBsAg and anti HBc tests on HBV reactivation; (3) whether host factors (DNA polymorphism) may help predict HBV reactivation. A larger patient cohort is needed to identify (1) baseline features that may help predict HBV reactivation, and (2) on-treatment features that may help timely anti-viral therapy.

DETAILED DESCRIPTION:
Treatment plan:

A typical course of rituximab-CHOP chemotherapy is as follows:

rituximab 375 mg/m2 i.v., day 1, cyclophosphamide 750 mg/m2 i.v., day 1, doxorubicin 50 mg/m2 i.v., day 1, vincristine 1.4 mg/m2 (maximal 2 mg) i.v., day 1, prednisolone 40 mg/m2/day p.o., day 1 to day 5.

Typically the treatment will be repeated every 3 weeks. If the patients cannot recover from chemotherapy-induced toxicity at the schedule time of the next course of treatment, modification of chemotherapy dosage or delay of chemotherapy administration will be done according to local treatment standard and will be recorded.

The use of component therapy or granulocyte colony-stimulating factor will be at the discretion of individual investigator.

Auxiliary medication, such as anti-emetics, will be given according to local treatment guidelines.

Statistical consideration:

1. Database Management Procedures

   Standard module for description of standard operation procedures for data processing to ensure quality and validity of the data.
2. Presentation of Efficacy and safety Endpoints

   2.1. The primary endpoint of this study is the incidence of HBV reactivation, defined by a greater than 10-fold increase, compared with previous nadir levels, of HBV DNA, during rituximab-CHOP chemotherapy and within 1 year after the last course of rituximab-CHOP chemotherapy.

   2.2. Secondary endpoints: Incidence of hepatitis , defined as a greater than 3 fold increase of serum ALT level that exceeded 100 IU/L.

   Incidence of severe hepatitis, defined as a hepatitis flare with an increase of ALT to more than 10 fold of ULN or bilirubin to more than 1.5 fold of ULN.

   Association between HBV reactivation and serological breakthrough (i.e., re-appearance of HBsAg) during follow-up Association between HBV reactivation and levels of anti-HBc antibodies during follow-up Association between HBV reactivation and HLA germline polymorphism (HLA-DPA1, HLA-DPB1, HLA-DQA1, HLA-DQB1, HLA-DRB1) / IL28B genotype of the patients Progression-free survival and overall survival for patients who receive rituximab-CHOP chemotherapy.
3. Hypotheses and Sample Size Determination

   It is estimated that in Taiwan the incidence of 'resolved' HBV infection in the general population is about 50%. A recent survey of HbsAg(-)blood donors indicated that 7% of the donors had detectable HBV DNA in serum. The incidence of diffuse large B-cell non-Hodgkin's lymphoma in Taiwan is 700-800 new patients/year (Taiwan Cancer Registry, http://crs.cph.ntu.edu.tw). We plan to enroll 150 patients in three years (50 new patients every year).
4. General Statistical considerations

   4.1 Randomization and stratification

   This is a single-arm study. No randomization will be done.

   4.2 Analysis population

   This study will enroll NHL patients with evidence of 'resolved' HBV infection. Eligible subjects must be negative for serum HBV surface antigen (HBsAg) and positive for at least one of the following in the serum: anti-core antigen (anti-HBc), anti-surface antigen (anti-HBs), or HBV DNA. Patients who receive at least 1 dose of rituximab-CHOP chemotherapy will be enrolled in to the intent-to-treat population and safety population. Patients who complete at least 1 course of rituximab-CHOP chemotherapy will be enrolled into the per-protocol analysis. The primary and secondary endpoints described in Section 2.1, 2.2, and 2.3 will be included in the per-protocol analysis.

   4.3 Dropout

   Taking into account 10% dropout rate, we need to enter 62 patients per year to the trial so that we may finish accrual of patients within 3 years.

   4.4 Baseline

   Before the first course of rituximab-CHOP chemotherapy, the baseline characteristics for each patient will be measured.

   4.5 Multicenter study

   This study will be conducted by all participating medical centers to the Lymphoma Disease Committee (14 centers in total). Since the rituximab-CHOP chemotherapy is the standard first-line treatment for patients with diffuse large B-cell NHL and follicular cell NHL, no center interaction on treatment is expected in this study.

   4.6 Adjustment for multiple testing

   Adjustment because of multiple testing is not needed in this study.

   4.7 Subgroup analysis

   Pre-specified subgroup analysis for the primary endpoint (HBV reactivation rate) will be done in the following sub-groups:
   1. baseline HBV DNA (+) vs. HBV DNA (-);
   2. baseline alanine transaminase (ALT) normal vs. abnormal.

   4.8 Patient Listings

   Individual patient listings should be also provided.
5. Interim analysis and data monitoring

   No interim analysis is planned for this study.
6. Final Analysis

For the final statistical analysis, this section should state the specific statistical procedures described in item 6 of this section in the analysis of every primary and secondary efficacy and safety endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diffuse large B-cell or follicular B-cell non-Hodgkin's lymphoma, for which chemotherapy with rituximab-CHOP chemotherapy is considered treatment-of-choice.
2. Evidence of 'resolved' HBV infection. Eligible subjects must be negative for serum HBV surface antigen (HBsAg) and positive for anti-core antibody (anti-HBc).
3. Age >18 years.
4. Performance status with ECOG score 0-2.
5. No previous chemotherapy and radiotherapy, no concurrent glucocorticoid use.
6. Absolute neutrophil count (ANC) > 1,500/mm3, platelet > 100,000/mm3 in the peripheral blood.
7. Total bilirubin < 2.5 mg/dl. Alanine aminotransferase (ALT) < 3 times UNL (upper limits of normal range).
8. Serum creatinine < 1.5 mg/dl. 9.10.Life expectancy 3 months.

11.Signed informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Patients with history of brain metastasis or CNS involvement.
3. Child's class B or C in patients with liver cirrhosis.
4. Impaired cardiac function with NYHA (New York Heart Association) classification Gr II.
5. History of other liver diseases such as hepatitis C, D, autoimmune hepatitis, primary biliary cirrhosis, Wilsons' disease.
6. Other major systemic disease, such as active infection, significant cardiac disease, neurological deficit or psychiatric disorder, that the investigators consider to be significant risk.
7. Any concomitant cancer treatment.
8. Known hypersensitivity of any of the study drugs (rituximab, cyclophosphamide, vincristine, doxorubicin, and prednisolone).
9. Known human immunodeficiency virus (HIV) infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
enroll 150 patients | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, Ph.D, Study Director — National Health Research Institutes, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No